CLINICAL TRIAL: NCT01218607
Title: BOsentan for Mild Pulmonary Vascular Disease in Asd Patients (the BOMPA Trial): a Double-blind, Randomized Controlled, Pilot Trial
Brief Title: Bosentan for Mild Pulmonary Vascular Disease in Asd Patients.
Acronym: BOMPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Alexander Van De Bruaene, Dr, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UZL-S52480
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Heart Septal Defects, Atrial
Keywords: Heart Septal Defects, Atrial; Pulmonary Circulation; Ventricular Function, Right; Echocardiography, Stress; Ergometry; Tissue Doppler Imaging
MeSH Terms: conditions — Heart Septal Defects, Atrial | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Active (Active Comparator)
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — Treatment will be initiated at a dose of 62.5 mg twice daily for 4 weeks and then increased to the maintenance dose of 125 mg twice daily for 12 weeks.
  Other Names: Bosentan = Tracleer
  Arms: Active
Drug: Placebo — Placebo will be taken twice daily for 16 weeks
  Arms: Placebo

SUMMARY:
Volume overload due to left-to-right shunting in patients with atrial septal defect type secundum causes pulmonary vascular disease over a long period of time. Pulmonary vascular resistance can be assessed non-invasively using bicycle stress echocardiography. By measuring cardiac output and pulmonary artery pressures at different stages of exercise, a pressure-output plot can be obtained. The slope of the pressure-output plot reflects pulmonary vascular resistance. In patients undergoing ASD repair after the age of 40 years, pulmonary vascular resistance was higher when compared to age-matched controls, indicating the presence of mild pulmonary vascular disease. Bosentan has been shown to decrease pulmonary vascular resistance.

The investigators hypothesize that in patients with an ASD type secundum, who underwent ASD repair after the age of 40 years, administration of bosentan decreases pulmonary vascular resistance as assessed by bicycle stress echocardiography.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   1.1 MEDICAL BACKGROUND

   Atrial septal defect (ASD) represents approximately 10% of all congenital heart diseases and is the third most common form of congenital heart defect. The incidence of congenital heart disease in Belgium is 1%, with ASD accounting for 25% of the cases (Data from the database of congenital heart diseases UZ Leuven.) Characterized by a free communication between the left and the right atrium, it may take the form of an ostium secundum defect (in the region of the fossa ovalis); an ostium primum defect (in the lower part of the atrial septum and associated with mitral regurgitation) or a sinus venosus defect (in the upper atrial septum and associated with anomalous drainage of one or more pulmonary veins)

   Patients with atrial septal defect (ASD) initially present with a left-to-right shunt, which may cause elevated pulmonary artery pressures at rest and/or during exercise. However, this persistently elevated pulmonary blood-flow also causes progressive lesions of the pulmonary vasculature, as first described by Heath and Edwards. The earlier stages present with medial hypertrophy and/or intimal proliferation and are largely reversible after closure of the defect. Later stages, however, are irriversible: the origin of pulmonary arterial hypertension (PAH). Eventually, this volume and pressure overload of the right heart may lead to heart failure and/or arrhythmias. As PVR exceeds systemic resistance, the shunt is reversed (right-to-left shunt) leading to systemic arterial desaturation (and the related consequences: polyglobulia, hyperuricemia, decreased renal function and abnormal coagulation): the Eisenmenger syndrome (ES). When occlusive fibrotic lesions have developed later in life, closure of the ASD, although still feasible, may not result in complete normalization of pulmonary artery pressures. Moreover, it has been shown that closure after the age of 40 years is associated with worse outcome. It has been suggested that an abnormal increase in pulmonary artery pressures during exercise reflects mild pulmonary vascular disease. However, pulmonary artery pressures are defined by both cardiac output and pulmonary vascular resistance. During exercise, the relationship between pulmonary artery pressures and cardiac output is slightly curvilinear because of a natural distensibility of the pulmonary arterioles. Using bicycle stress echocardiography, pulmonary vascular resistance can be estimated either as a ratio of pulmonary artery pressure and cardiac output at each stage (total PVR) or by using linear regression analysis of the pressure-flow plots (dynamic PVR).

   Prognosis of patients with unrepaired ASDs is thought to be shortened and repair can avoid right ventricular (RV) failure, pulmonary hypertension, thrombo-embolic events and atrial dysrrhythmias. So, when the defect is discovered early, an ASD is usually closed in childhood, unless the defect is considered not to be clinical significant. Sometimes, as most patients with an isolated ASD are asymptomatic during childhood, an ASD comes to medical attention at an older age.

   Patients with a corrected ASD have a poorer prognosis than patients in a control group, especially in the presence of PAH, which confers an eightfold increased probability of functional limitations. In the Euroheart survey PAH was present in 12% of patients with a closed ASD. As PAH is a progressive disease, early diagnosis and treatment may improve outcome in these patients.

   A first analysis of data obtained from the registry of ASD showed that in the transcatheter closed ASD patients, mPAP was the only independent predictor of atrial arrhythmia after ASD repair. Moreover, our first prospective study showed that it is possible to identify patients with mild pulmonary vascular disease using stress echocardiography and that patients with an ASD closed at later age were unable to decrease pulmonary vascular resistance during exercise, resulting in a higher pulmonary vascular resistance at peak exercise when compared to a control group. This was reflected in a steeper pressure-flow plot when compared to healthy controls. Endothelin has shown to influence vasomotor tone, especially during exercise. Moreover, Faoro et al showed that bosentan decreased pulmonary vascular resistance as assessed with pressure-flow plots during hypoxia. Therefore, this study was designed to evaluate the effect of an dual endothelin receptor antagonist on total pulmonary vascular resistance during exercise in an older ASD patient population.

   1.2 DRUG PROFILE

   Mechanism of action

   Bosentan is a dual endothelin receptor antagonist (ERA) with affinity for both endothelin A and B (ET-A and ET-B) receptors. Bosentan decreases both pulmonary and systemic vascular resistance resulting in increased cardiac output without increasing heart rate.

   The neurohormone endothelin-1 (ET-1) is one of the most potent vasoconstrictors known and can also promote fibrosis, cell proliferation, cardiac hypertrophy, and remodeling and is pro-inflammatory. These effects are mediated by endothelin binding to ET-A and ET-B receptors located in the endothelium and vascular smooth muscle cells. ET-1 concentrations in tissues and plasma are increased in several cardiovascular disorders and connective tissue diseases, including pulmonary arterial hypertension, scleroderma, acute and chronic heart failure, myocardial ischaemia, systemic hypertension and atherosclerosis, suggesting a pathogenic role of ET-1 in these diseases. In pulmonary arterial hypertension and heart failure, in the absence of endothelin receptor antagonism, elevated ET-1 concentrations are strongly correlated with the severity and prognosis of these diseases.

   Bosentan competes with the binding of ET-1 and other ET peptides to both ET-A and ET-B receptors, with a slightly higher affinity for ET-A receptors (Ki = 4.1-43 nM) than for ET-B receptors (Ki = 38-730 nM). Bosentan specifically antagonises ET receptors and does not bind to other receptors.

   1.3 RATIONALE FOR PERFORMING THE STUDY

   Although an ASD seems an easily correctable defect, patients with a repaired ASD have a poorer prognosis than patients in a control group, especially in the presence of PAH, which confers an eightfold increased probability of functional limitations. In the Euroheart survey PAH was present in 12% of patients with a closed ASD. Whether it is useful to treat mild to moderate pulmonary vascular disease after repair of an ASD with specific PAH treatment in order to have a positive effect on exercise capacity and even outcome outcome still needs to be evaluated.

   As outlined in section 1.1, the investigators were able to identify patients with mild pulmonary vascular disease using bicycle exercise echocardiography. Patients with an ASD repaired after the age of 40 years appeared to have higher PVR when compared to healthy controls. Moreover, in older patients a higher mPAP at diagnosis was an independent predictor for the occurrence of late atrial arrhythmias.

   Therefore, the present study will investigate whether bosentan has a beneficial effect on PVR as measured with bicycle stress echocardiography in patients with repaired ASD and WHO FC II mild pulmonary vascular disease using dynamic PVR as a surrogate endpoint.

   1.3.1 DOSE AND POSOLOGY

   Treatment will be initiated at a dose of 62.5 mg twice daily for 4 weeks and then increased to the maintenance dose of 125 mg twice daily for 12 weeks.

   Dosage in elderly patients: No dosage adjustment in required in patients over the age of 65 years.
2. STUDY OBJECTIVES

   The primary efficacy objective is to assess the efficacy of the dual active endothelin receptor antagonist bosentan in patients with WHO functional class II mild to moderate PAH after surgical or interventional closure of an ASD .
3. STUDY DESIGN

This is a prospective, monocentric, randomised, double-blind, placebo-controlled, pilot study to evaluate the efficacy of dual active endothelin receptor antagonist bosentan in patients with WHO FC II, mild pulmonary vascular disease after ASD repair.

4 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

The null hypothesis of the study is that in patients receiving specific PAH treatment no change in PVR is observed. This trial aims to demonstrate to efficacy of bosentan to lower PVR as assessed by bicycle exercise echocardiography in patients with surgically or transcatheter closed ASD.

5 RANDOMISATION

Patients will be randomly assigned to treatment groups with equal probability of assignment to each treatment arm (allocation ratio 1:1). The randomisation schedule will be generated using validated software. The investigators will remain blinded to the randomisation schedule until after the final database is locked. The randomisation schedule will be examined only if required by an emergency. Any such break should be documented clearly.

6 SAMPLE SIZE CALCULATION

As the study design is considered as a pilot trial, it primarily aims at defining means and standard deviations in both treatment arms in order to allow for future sample size calculations.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by patient prior to initiation of any study-mandated procedure.
* Male or female patients > 40 years with atrial septal defect type secundum and > 40 years of age at the time of repair
* Women of childbearing potential must have a negative pre-treatment pregnancy test and must use a reliable method of contraception during study treatment and for at least 3 months after study treatment termination.
* Women not of childbearing potential are defined as postmenopausal (amenorrhea for at least 1 year), or documented surgically or naturally sterile.

Exclusion Criteria:

* Pregnancy or lactation
* Women of child-bearing age who are sexually active without practising reliable methods of contraception
* Any disease or impairment that, in the opinion of the investigator, excludes a subject from participation
* Substance abuse (alcohol, medicines, drugs)
* Other medical, psychological or social circumstances that would adversely affect a patient's ability to participate adequately in the study or increase the risk to the patient or others in the case of participation
* Insufficient compliance
* Subjects who are not able to perform cardiopulmonary exercise testing
* ASD repair < 6 months before inclusion
* PAH of any aetiology other than the one specified in the inclusion criteria
* Impairment of organic function (renal, hepatic)
* Arterial hypotension (systolic blood pressure < 85 mmHg)
* Anaemia (Hb< 10 g/dl)
* Decompensated symptomatic polycythemia
* Thrombocytopenia (< 50000/µl)
* Significant valvular diseases, other than tricuspid or pulmonary regurgitation
* Chronic lung disease or total lung capacity < 80% of predicted value
* History of significant pulmonary embolism
* Other relevant diseases (HIV infection, Hep B/C infection)
* Subjects with known intolerance to bosentan or their constituents
* Prohibited medication: any medication listed below which has not been discontinued at least 30 days prior to screening

  * Unspecified or other significant medication (glyburide or immunosuppression)
  * Drugs to treat PAH (endothelin receptor antagonists, PDE-5 antagonists, prostanoids)
  * Medication that is not compatible with bosentan or that interferes with its metabolism (inhibitors of CYP2C9 or CYP3A4) or that, in the investigator's opinion, may interfere with bosentan treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary vascular resistance | 16 weeks
  Pulmonary vascular resistance can be measured using bicycle stress echocardiography by estimating the slope of a pressure-flow plot using linear regression analysis.

SECONDARY OUTCOMES:
Peak oxygen consumption | 16 weeks
  The highest oxygen uptake available by bicycle ergometry despite further work rate increases and effort by the subject.
Right ventricular function | 16 weeks
  Right ventricular function as assessed by echocardiography.
Liver function abnormalities | 4, 8,12 and16 weeks
  An increase in ASAT and/or ALAT equal or more than 3 times the upper limit of normal.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Budts, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium